CLINICAL TRIAL: NCT06606262
Title: Tonsillectomy Versus Tonsillotomy in the Treatment of Recurrent Acute Tonsillitis: A Randomized Controlled Non-inferiority Trial
Brief Title: Tonsillectomy Versus Tonsillotomy in the Treatment of Recurrent Acute Tonsillitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tejs Ehlers Klug (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Sponsor-Investigator, Tejs Ehlers Klug, MD, DMSc, Clinical Associate Professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TETO study protocol
Record Dates: First submitted 2024-08-26; First posted 2024-09-20 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Tonsillitis Recurrent
Keywords: tonsillectomy; tonsillotomy; quality of life
MeSH Terms: interventions — Tonsillectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tonsillotomy (Experimental): A potential non-inferior surgical procedure for treating recurrent acute tonsillitis.
  Interventions: Procedure: Tonsillotomy
- Tonsillectomy (Active Comparator): The current standard surgical procedure for treating recurrent acute tonsillitis.
  Interventions: Procedure: Tonsillectomy

INTERVENTIONS:
Procedure: Tonsillotomy — Bilateral partial removal of the palatine tonsils to a level between the pharyngeal pillars and the tonsillar capsule. Surgery will be performed under general anesthesia using monopolar electrocautery.
  Other Names: Intracapsular tonsillectomy; TO
  Arms: Tonsillotomy
Procedure: Tonsillectomy — Bilateral extracapsular removal of palatine tonsils. Surgery will be performed under general anesthesia using "cold knife" dissection.
  Other Names: Extracapsular tonsillectomy; TE
  Arms: Tonsillectomy

SUMMARY:
Background: recurrent acute tonsillitis (RT) is a frequent condition affecting teenagers and adults. Patients suffer from recurring throat symptoms, fever and impaired quality of life (QOL). Tonsillectomy (TE) is the only well-known treatment, but studies indicate that tonsillotomy (TO) is associated with less morbidity (eg. pain and bleeding) and equal efficiency (e.g. reduced number of sore throat episodes and improved QOL). The investigator aim to clarify whether TO is a non-inferior alternative to TE.

Methods: inclusion and randomization of 250 adult RT patients for TE or TO with a 12 month follow up. Comparisons will be made between groups, and outcome measures includes number of sore throat episodes, QOL and postoperative pain.

Discussion: the study has the potential to improve the treatment of a prevalent disease by enhancing knowledge of an alternative procedure (TO) associated with less discomfort and risk than the current standard procedure (TE) and a presumably low risk of insufficiency.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥15 years) with RT, defined as a minimum of five tonsillitis episodes in one year or a minimum of three tonsillitis episodes per year for two years (Danish National Guidelines criteria
* The ability to understand Danish orally and in writing.

Exclusion Criteria:

* Previous TE or TO.
* Suspected tonsillar malignancy.
* History of malignant tumor in the oral cavity, the pharynx or the larynx.
* Previous radiation therapy on head or neck.
* Hemorrhagic diathesis or anticoagulant therapy.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of sore throat episodes after TE vs. TO. | 12 months (and 24, 36 and 60 months)
QOL measured as postoperative Tonsillectomy Outcome Inventory 14 (TOI-14) score after TE vs. TO | 12 months (and 24, 36 and 60 months)
  A disease-specific questionnaire for adults with tonsillitis. It is used pre- and postoperatively to detect changes in quality of life. It consists of 14 questions that covers four subscales: throat dis-comfort (question 1-4) general health (question 5-6), resources (question 7-10), and social psychological restrictions (question 11-14). The questionnaire uses a six-point Likert scale with 0 representing "no problem" and 5 representing "couldn't be worse". The points are summed, divided by the number of questions multiplied by 5, and multiplied by 100, giving scores in the range 0-100, where higher scores reflect poorer quality of life
Summarized postoperative pain scores (days 1-10) | Days 1-10
  Measured on a numeric rating scale from 0 til 10 in which 0 represents "no pain" and 10 represents "excruciating pain"
Overall postoperative discomfort (day 21) | Day 21
  Measured on a numeric rating scale from 0 til 10 in which 0 represents "no discomfort" and 10 represents "excruciating discomfort"

SECONDARY OUTCOMES:
Proportion of patients cured (defined as postoperative TOI-14<15) after TE vs. TO | 12 months (and 24, 36 and 60 months)
Overall patient satisfaction after TE vs. TO | 12 months (and 24, 36 and 60 months)
  Patients will be asked the following question: "Keeping in mind your full experience and the effects of surgery so far, are you satisfied with having undergone surgery?. Possible answers are 1) "yes", 2) "no" and 3) "I don't know"
Postoperative Glasgow Benefit Inventory (GBI) score after TE vs. TO | 12 months (and 24, 36 and 60 months)
  A generic questionnaire for otorhinolaryngological interventions. It is used post-intervention to detect changes in quality of life. It consists of 18 questions that covers three subscales: a general health sub-scale (question 1-6, 9-10, 14, 16-18), a social support subscale (question 7, 11 and 15) and a physical health subscale (question 8, 12-13). The questionnaire uses a five-point Likert scale with 1 representing "worst change of health status" and 5 representing "best change of health status". The points are summed and divided by the number of questions (resulting in average scores), and by subtracting 3 and multiplying by 50, the final scores range from -100 to +100. 0 indicates no change, higher scores reflect better quality of life
Number of sore throat days after TE vs. TO | 12 months (and 24, 36 and 60 months)
Prevalence of reoperation after TE vs. TO | 12 months (and 24, 36 and 60 months)

CONTACTS AND LOCATIONS:
Locations (2):
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-19): https://cdn.clinicaltrials.gov/large-docs/62/NCT06606262/Prot_SAP_000.pdf